CLINICAL TRIAL: NCT05868148
Title: Shoulder iD™ Primary Reversed Glenoid Outcomes Clinical Study
Acronym: SiD
Status: Active, not recruiting | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: UE-02-2021
Record Dates: First submitted 2023-04-21; First posted 2023-05-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff Tears; Rheumatoid Arthritis Shoulder; Osteoarthritis Shoulder; Avascular Necrosis of the Head of Humerus; Fracture, Humeral; Traumatic Arthritis of Right Shoulder Region (Diagnosis); Shoulder Deformity
Keywords: Massive RCT; Non-repairable RCT; Glenohumeral joint
MeSH Terms: conditions — Rotator Cuff Injuries; Humeral Fractures; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Shoulder iD device implant: Adult patients who have reached skeletal maturity, with a functional deltoid muscle, and massive and non-repairable rotator cuff tear within one or more indications and zero contraindications who will receive the Shoulder iD Primary Reversed Glenoid device to replace the shoulder joint.
  Interventions: Device: Shoulder iD™ Primary Reversed Glenoid

INTERVENTIONS:
Device: Shoulder iD™ Primary Reversed Glenoid — Device implant via reversed total shoulder arthroplasty
  Other Names: Patient-Matched Primary Reversed Glenoid

SUMMARY:
The goal of the Shoulder iD™ Primary Reversed Glenoid Outcomes Clinical Study is to collect safety and performance data on the commercially available Shoulder iD™ Primary Reversed Glenoid device. The study will learn about standard device use in adult patients who have a functional deltoid muscle and massive and non-repairable rotator cuff tear. The main questions it aims to answer are:

* What is the average improvement in patient-reported shoulder function after 2 years when compared to before the surgery, and
* What is the rate of surgical revisions needed over a 10 year period

Patients will be asked to will be asked to regularly attend their check-up visits with their surgeon (including having x-rays or CT images taken to check their shoulder and implant), to complete questionnaires to report how their shoulder is doing, and to tell their surgeon when they notice any changes.

DETAILED DESCRIPTION:
The Shoulder iD™ Primary Reversed Glenoid Outcomes Clinical Study is a Global, single arm, multicenter, prospective, non-significant risk Post-Market Clinical Follow-up (PMCF) study, designed to collect safety and performance data on designated commercially available Shoulder iD™ Primary Reversed Glenoid.

The objective of this multicenter study is to collect clinical data at baseline, surgery, immediate post-op, and annually through 10 years post-operation, on related clinical complications and clinical outcomes of market-approved Shoulder iD™ Primary Reversed Glenoid, to demonstrate safety and performance of these implants in a real-world setting.

The primary outcome measure is the average improvement in American Shoulder and Elbow Surgeons (ASES) score from baseline to 24 months.

Secondary outcome measures include the following assessments to be evaluated throughout the patient's participation in the study:

* Constant Score (years 1, 2, 5 and 10 only)
* Single Assessment Numeric Evaluation (SANE) Score
* Patient Satisfaction
* EQ-5D-5L

Radiologic imaging: Patient images (X-ray or CT) completed at baseline and in-person follow-ups will be analyzed for standard radiographic findings, including, but not limited to: device migration, component breakage, radiolucencies and bone characteristics.

Revision rate and survivorship will be assessed annually and at any time upon request for regulatory purposes such as PMCF or Clinical Evaluation Report (CER) updates. The cumulative incidence of device revisions and reoperations will be reported as well as Kaplan-Meier estimates for implant survival.

Adverse events will be evaluated from inclusion to last follow-up and will be documented during the study and categorized as whether they are serious and whether they are related to the Sponsor device or implant procedure.

During the study, patients will undergo the following procedures, which are standard of care:

* Patient information and Consent (as applicable per local regulation),
* Inclusion/non-inclusion criteria,
* Demography, Height & Weight,
* Surgical history and relevant medical history,
* Physician exams (Range of Motion and Strength measurements),
* Patient questionnaires (ASES, Constant, SANE, Patient Satisfaction, EQ-5D-5L),
* Shoulder study implant & surgery related data,
* CT scans, x-rays
* AE / SAE collection (continuous recording).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of the informed consent or non-opposition (when applicable).
* Informed and willing to sign an informed consent form approved by IRB or EC (when applicable).
* Willing and able to comply with the requirements of the study protocol.
* Considered a candidate for shoulder arthroplasty using a study device.
* Meets indications for use requirements or other local, regional, or geographic specific regulatory requirements

Exclusion Criteria:

* Patients who are not able to comply with the study procedures based on the judgment of the assessor (e.g., cannot comprehend study questions, inability to keep scheduled assessment times).
* Patient belongs to a vulnerable group of patients, including minor patients, those unable to decide for themselves to participate or needing a Legally Authorized Representative (LAR), or others who could be subject to coercion (patients who may not be acting on their own initiative) (referred to as a "vulnerable subject" in section 3.44 of the ISO 14155:2020).
* Active local or systemic infection, sepsis, or osteomyelitis
* Poor bone quality, where there could be considerable migration of the prothesis and/or a chance of fracture of the humerus or glenoid (reassessed at time of surgery)
* Significant injury to the brachial plexus
* Inadequate bone stock in the proximal humerus or glenoid fossa for supporting the device components
* Neuromuscular disease (e.g., joint neuropathy) Known allergy to one of the product materials
* Metabolic disorders which may impair bone formation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intended patient population are adult patients who have reached skeletal maturity, with a functional deltoid muscle, and massive and non-repairable rotator cuff tear within one or more indications and zero contraindications with pain disabled by:
  * Rheumatoid arthritis
  * Non-inflammatory degenerative joint disease (i.e. osteoarthritis and avascular necrosis)
  * Correction of functional deformity
  * Fractures of the humeral head
  * Traumatic arthritis
  * Revision of glenohumeral joint if sufficient native glenoid bone remains
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Performance: change in functional ability of the treated shoulder | from baseline to 24 months
  The average change in functional ability as measured by the American Shoulder and Elbow Surgeons (ASES) score. ASES is an absolute score ranging from 0 to 100 where a higher score indicates better shoulder function.
Safety: Revision rate and device survivorship | from date of inclusion until date of study exit (study completion or early termination for any cause), assessed up to 10 years
  The cumulative incidence of device revisions and reoperations

SECONDARY OUTCOMES:
Performance: change in level of pain and ability to carry out normal daily activities of the patient | from date of inclusion until date of study exit (study completion or early termination for any cause), assessed up to 10 years
  Assessed via the Constant-Murley Shoulder score collected at baseline, years 1, 2, 5 and 10 and any other standard collection timepoint. In this score, 35 points are allocated for subjective assessments of pain and activities of daily living and 65 points are available for objective measures of rage of movement and shoulder strength. A score of 100 is a healthy shoulder.
Performance: change in patient self-assessment of current status of their treated shoulder | from date of inclusion until date of study exit (study completion or early termination for any cause), assessed up to 10 years
  Assessed via the Single Assessment Numeric Evaluation (SANE) score collected from patients via ePRO at baseline, 3 months, and annually. The rating is from 0% to 100% with 100% being normal.
Performance: change in patient self-rated quality of life | from date of inclusion until date of study exit (study completion or early termination for any cause), assessed up to 10 years
  Assessed via EQ-5D-5L Five Dimensions Quality of Life measurement general health questionnaire collected from patients via ePRO at baseline, 3 months and annually. Each dimension is measured on 5 levels from 1 being no problems to 5 being extreme problems.
Performance: change in patient satisfaction with their shoulder | from date of inclusion until date of study exit (study completion or early termination for any cause), assessed up to 10 years
  Satisfaction rating collected from patients via ePRO at baseline, 3 months and annually. Rating options are: Very Satisfied, Satisfied, Dissatisfied, and Very Dissatisfied.
Safety: Adverse Event rate and assessments | from date of treatment until date of study exit (study completion or early termination for any cause), assessed up to 10 years
  Cumulative incidence of procedure and/or device related events (ADE, AESI, SAE, SADE)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma and Extremities
Locations (5):
- United States (5):
  - UCSF, San Francisco, California
  - Jameson Crane Sports Medicine Institute OSU, Columbus, Ohio
  - UT Southwestern, Frisco, Texas
  - UT Health Science center - Houston, Houston, Texas
  - Carilion Clinic, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No